CLINICAL TRIAL: NCT07399756
Title: Assessment of Mitochondrial Parameters in Blood Before and After S-Ketamine Treatment
Brief Title: Mitochondrial Function After Ketamine
Status: Not yet recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-05-2419-RA-CTIL
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: ketamine, Mitochondrial, Treatment-Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mitochondrial DNA (mtDNA) copy number will be assessed using quantitative real-time PCR (RT-qPCR) from DNA isolated from PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ketamine inhalation group: Treatment-Resistant Depression patient after Ketamine inhalation
  Interventions: Drug: S (+) Ketamine

INTERVENTIONS:
Drug: S (+) Ketamine — the patients are treated with S-Ketamine in order to treat there Treatment-Resistant Depression via inhalation

SUMMARY:
The goal of this observational study is to learn about the role of mitochondria in response to S-ketamine. in individuals with Treatment-Resistant Depression.

the Research Questions are

1. Does S-ketamine treatment modulate mitochondrial function in peripheral blood cells, as reflected by mitochondrial content and circulating mitochondrial biomarkers such as GDF15?
2. Can changes in mitochondrial function serve as biomarkers for predicting or monitoring clinical response to S-ketamine treatment?

Samples will be collected at baseline, 3 hours after the first treatment, and 6 weeks post-exposure, and compared between responders and non-responders

ELIGIBILITY:
Inclusion Criteria:

Male or female, 18-65 years of age Diagnosis of Major Depressive Disorder according to the DSM-V Patient has a HAM-D≥23 Treatment resistant -Did not respond to two antidepressants trial Medically stable: No active physical disease: malignancy, cardiac condition, hypertension , stable medications for the past month etc.

Exclusion Criteria:

Known sensitivity to ketamine drug or alcohol abuse Patient taking lithium or corticosteroids Pregnant or breast-feeding has another axis I diagnosis attention deficits disorder a history or current serious neurological, metabolic autoimmune bone marrow, oncologic or additional psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit ten normal controls, 30 Patients with the diagnosis of treatment-resistant depression (TRD), failed to at least two antidepressants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
S-ketamine effects on the mitochondrial | 3 hours and 6 weeks
  Does S-ketamine treatment modulate mitochondrial function in peripheral blood cells, as reflected by mitochondrial content and circulating mitochondrial biomarkers such as GDF15?

OTHER OUTCOMES:
mitochondrial function as a biomarker for S-ketamine treatment | 3 hours and 6 weeks
  Can changes in mitochondrial function serve as biomarkers for predicting or monitoring clinical response to S-ketamine treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel